CLINICAL TRIAL: NCT04194060
Title: Enhanced Recovery After Surgery Versus Conventional Approach in Peptic Perforation-A Randomized Control Trial
Brief Title: ERAS vs Conventional Approach in Peptic Perforation-RCT
Acronym: ERASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Tushar Subhadarshan Mishra, Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIIMS BBSR/PGT/2019-20/65
Record Dates: First submitted 2019-11-22; First posted 2019-12-11 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Peptic Ulcer Perforation; Perforated Bowel; Post-Op Complication; Emergencies; Perioperative Complication
Keywords: ERAS; Emergency surgery; Fast track surgery; Perioperative Care; Enhanced recovery after surgery
MeSH Terms: conditions — Peptic Ulcer Perforation; Intestinal Perforation; Postoperative Complications; Emergencies | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patient will be allocated into two arms, ERAS(Enhanced recovery after surgery) group and Conventional group. 30 patients will be recruited in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced recovery after surgery group (Experimental): ERAS GROUP
  * Tracheal intubation.
  * Short acting anesthetic agents,avoid opioid agents
  * Omental patch repair with placement of sub hepatic drain
  * Bilateral Transverse abdominis plane block/ Rectus sheath block immediately after surgery.
  * Post operative nausea and vomiting prophylaxis.
  * Encourage to mobilize out of bed after effect of general anesthesia has weaned off.
  * Initiation of feeding-Oral sips on day 1, step up day 2 onward
  * Removal of nasogastric tube-immediately after surgery after aspirating the gastric content through nasogastric tube.
  * Removal of urinary catheter-after weaning from the effect of general anesthesia.
  * Sub hepatic drain removal -anytime within 24 hours;drain will not be removed if fluid is bilious or pus.
  * Avoid opiod analgesics.
  Interventions: Combination Product: Enhanced Recovery after Surgery group
- Conventional group (Active Comparator): CONVENTIONAL GROUP
  * Tracheal intubation
  * Short acting anesthetic agents, avoid opiod anesthesia agents.
  * Omental patch repair along with sub hepatic drain placement.
  * Post operative nausea and vomiting prophylaxis.
  * Ambulation-as per patients' own request.
  * Initiation of oral feed- after passage of 1st flatus.
  * Nasogastric tube removal-output <300ml/day with resolution of ileus.
  * Removal of urinary catheter- when patient sits on bed side/ambulate.
  * Removal of sub hepatic drain-when patient tolerates unrestricted amount of liquid diet and drain output is less than 200 ml /day.
  * Patient will receive opiod analgesics.
  I
  Interventions: Combination Product: Conventional

INTERVENTIONS:
Combination Product: Enhanced Recovery after Surgery group — * Tracheal intubation and with General anesthesia
  * Short acting anesthetic agents,avoid opioid agents
  * Omental patch repair with placement of sub hepatic drain
  * Bilateral Transverse abdominis plane block/ Rectus sheath block immediately after surgery.
  * Post operative nausea and vomiting prophylaxis.
  * Encourage to mobilize out of bed after effect of general anesthesia has weaned off.
  * Initiation of feeding-Oral sips on day 1, step up day 2 onward
  * Removal of nasogastric tube-immediately after surgery after aspirating the gastric content through nasogastric tube.
  * Removal of urinary catheter-after weaning from the effect of general anesthesia.
  * Sub hepatic drain removal -anytime within 24 hours;drain will not be removed if fluid is bilious or pus.
  * Avoid opiod analgesics.
  Arms: Enhanced recovery after surgery group
Combination Product: Conventional — Tracheal intubation
  * Short acting anesthetic agents, avoid opiod anesthesia agents.
  * Omental patch repair along with sub hepatic drain placement.
  * Post operative nausea and vomiting prophylaxis.
  * Ambulation-as per patients' own request.
  * Initiation of oral feed- after passage of 1st flatus.
  * Nasogastric tube removal-output <300ml/day with resolution of ileus.
  * Removal of urinary catheter- when patient sits on bed side/ambulate.
  * Removal of sub hepatic drain-when patient tolerates unrestricted amount of liquid diet and drain output is less than 200 ml /day.
  * Patient will receive opiod analgesics.
  Arms: Conventional group

SUMMARY:
This study compares 2 different ways of perioperative management in patients of peptic perforation. Experimental arm is the ERAS arm( Enhanced recovery after surgery) and the comparative arm is Conventional arm.

DETAILED DESCRIPTION:
While the conventional approach to perioperative management can potentially prolong the post operative hospital stay, ERAS(Enhanced recovery after surgery), a multi-modal and multispeciality approach to perioperative management may reduce the length of hospital stay. In the preoperative period, patients will be counselled regarding the operative procedure and particulars of the perioperative management.In the intra-operative period short acting general anesthetic agents and short acting muscle relaxants will be used.Intravenous fluid administration will be goal directed. After the operative procedure, bilateral rectus sheath block will be administered. Patient will also receive post-operative nausea and vomiting prophylaxis. Nasogastric tube will be removed immediately after the operative procedure. In the post operative period, patients will be encouraged to ambulate early. Enteral nutrition will be initiated as early as possible. Indwelling catheters will be removed in the early post-operative procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with peptic perforation intra -operatively
2. Perforation of size <=1 cm
3. Patient age more than 18 years
4. American Society of Anesthesiologists score of I or II

Exclusion Criteria:

1. Refractory septic shock at presentation.
2. Known Chronic kidney disease/ Chronic liver disease patients
3. Pregnant patients.
4. Patients with history of chronic steroid abuse.
5. Intraoperatively

   * Patient with coexistent peptic perforation with bleeding ulcer.
   * Peptic perforation requiring procedure other than Omental patch repair.
   * Sealed perforations.
   * Malignant perforation.
6. Patient requiring Positive Pressure Ventilator support post operatively for more than 12 hours.
7. Patient requiring urinary catheterization for other indications.
8. Coexistent neurological or psychiatric illness or unable to understand the study.
9. Patient refusing for consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Post operative period up-to one month.
  Duration from the time of operation to time of discharge

SECONDARY OUTCOMES:
Recovery of functional parameters | Post operative period up-to one month.
  * Time of withdrawal of nasogastric tube (hours)
  * Time to first bowel sound (hours)
  * Time to first flatus (hours)
  * Time to first stool (hours)
  * Time to removal of drain(hours)
  * Time to first fluid diet (hours)
  * Time to first solid diet (hours)
  * Time to stoppage of IV fluids(hours)
  * Time of removal of urinary catheter (hours)
  * Time to ambulation(hours)
Post operative complications | Post operative period up-to three months.
  * Anastomotic leakage
  * Pneumonia
  * Ileus
  * Obstruction
  * Wound infection
  * Abdominal sepsis
  * Burst Abdomen
  * Need for reinsertion of nasogastric tube
  * Need for reinsertion of urinary catheter
  * Need for drainage of abdominal collection
  * Readmission
  * Re operation
  * Mortality

OTHER OUTCOMES:
Quality of life scoring and assessment | Post operative period - at day of discharge, at one month follow up and at third month follow up.
  Quality of life assessment will be done using EQ-5D-5L questionnaire (Euroqol 5 dimensions and 5 levels). It has 2 components, descriptive and objective. Descriptive component comprises of 5 dimensions which are mobility, self care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, namely no problem, slight problems, moderate problems, severe problems and extreme problems. Objective component is also called Euroqol visual analog scale. Score ranges from zero to hundred.The endpoints are labelled as 'the best health participant can imagine' and 'the worst health participant can imagine'. It will be assessed on the day of discharge, follow up at one month and follow up at third month in the post operative period.
Intra-abdominal collection | Post operative period-at one month and at third month in post operative period.
  Ultrasonography abdomen will be done at one month to look for any intra-abdominal collection and if any collection is found, will be repeated at third month follow up.
Hematological parameter | Post-operative period up-at one month and at third month.
  Total leukocyte count will be measured at follow up at one month.If the value is more than 11,000 cells/mm cube or less than 4000 cells/mm cube, then it will be measured again at third month of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: TUSHAR S MISHRA, MBBS,MS, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Tushar S Mishra, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohsina S, Shanmugam D, Sureshkumar S, Kundra P, Mahalakshmy T, Kate V. Adapted ERAS Pathway vs. Standard Care in Patients with Perforated Duodenal Ulcer-a Randomized Controlled Trial. J Gastrointest Surg. 2018 Jan;22(1):107-116. doi: 10.1007/s11605-017-3474-2. Epub 2017 Jun 26. PMID 28653239
- [Background] Lohsiriwat V, Jitmungngan R. Enhanced recovery after surgery in emergency colorectal surgery: Review of literature and current practices. World J Gastrointest Surg. 2019 Feb 27;11(2):41-52. doi: 10.4240/wjgs.v11.i2.41. PMID 30842811
- [Background] Agarwal A, Jain S, Meena LN, Jain SA, Agarwal L. Validation of Boey's score in predicting morbidity and mortality in peptic perforation peritonitis in Northwestern India. Trop Gastroenterol. 2015 Oct-Dec;36(4):256-60. doi: 10.7869/tg.300. PMID 27509704
- [Result] Gonenc M, Dural AC, Celik F, Akarsu C, Kocatas A, Kalayci MU, Dogan Y, Alis H. Enhanced postoperative recovery pathways in emergency surgery: a randomised controlled clinical trial. Am J Surg. 2014 Jun;207(6):807-14. doi: 10.1016/j.amjsurg.2013.07.025. Epub 2013 Oct 10. PMID 24119887